CLINICAL TRIAL: NCT06373679
Title: Non-cigarette Tobacco Products as Harm Reduction Tools in Smokers Who Failed to Quit With Traditional Methods
Brief Title: Switch or Quit R01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tracy Smith, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00125514; 1R01DA056445-01A1 (NIH)
Record Dates: First submitted 2024-04-05; First posted 2024-04-18 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cigarette Smoking; Smoking Behaviors
MeSH Terms: conditions — Cigarette Smoking; Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Choice of Medication (Experimental): This arm includes participants randomly assigned to the Meds Group. Participants will choose between 1) combo NRT and 2) varenicline. The NRT will consist of transdermal NRT and nicotine lozenge. Participants will receive study product for 11 weeks.
  Interventions: Behavioral: Switching using Medication
- Choice of E-Cigarette (Experimental): This arm includes participants randomly assigned to the E-Cigarette Group. Participants will choose between two different brands of e-cigarettes and choose up to two different flavors. Participants will receive study product for 11 weeks.
  Interventions: Behavioral: Switching to E-Cigarette

INTERVENTIONS:
Behavioral: Switching to E-Cigarette — Participants will receive eleven weeks of e-cigarette products with instructions to switch completely at switch date
  Arms: Choice of E-Cigarette
Behavioral: Switching using Medication — Participants will receive eleven weeks of FDA approved medication, either varenicline or combination NRT, with instructions to quit smoking cigarettes at quit date
  Arms: Choice of Medication

SUMMARY:
This study evaluates whether non-cigarette tobacco products (e-cigarettes) can help smokers quit smoking as compared to traditional quit methods (nicotine replacement therapy or varenicline/Chantix). Participants in this study will be randomly assigned to one of two groups, then will have a choice between the offered products of that group. Participants in the e-cigarette group will have a choice of e-cigarette brand and flavor. Participants in the medication group will have choice between nicotine replacement therapy (patches and lozenges) or varenicline, also known as Chantix. Participation will last 6 months and will include weekly phone calls for the initial 7-weeks plus a 11-week phone call and a 6-month follow-up visit. Participants will also complete electronic daily diaries during the first 7-weeks.

DETAILED DESCRIPTION:
Even though e-cigarettes have risen in prevalence over the last decade, data on the use of these products as harm reduction tools for smokers who try to switch completely is lacking.

These data are urgently needed for several reasons.

1. Clinicians cannot provide clear guidance to smokers who may be interested in switching. Questions from medical patients about e-cigarettes are on the rise, and data show that medical providers are providing mixed messages about the safety and utility of e-cigarettes, with some physicians discouraging their use and some recommending them as cessation aids.
2. Public health organizations are also providing mixed messages about the health risks of non-cigarette tobacco products-with some not recommending their use at all (The American Cancer Society, American Lung Association), and some acknowledging that complete switching to e-cigarettes would reduce health risks compared to continued smoking, but not recommending the use of these products over traditional methods (Centers for Disease Control, Food and Drug Administration).
3. In the absence of clear messaging about non-cigarette products, smokers who fail with traditional methods are continuing to smoke cigarettes, the most harmful tobacco product available.

The reviews underscore the need for additional data on this topic, especially data comparing the products to pharmacotherapy. The goal of the proposed study is to provide one of the first well-designed randomized controlled trials that addresses whether alternative tobacco products (e-cigarettes) have the potential to serve as harm reduction tools in a critical population-smokers who have tried to quit smoking using FDA-approved pharmacotherapy and failed to do so.

ELIGIBILITY:
Inclusion Criteria

* Adults 21+ who previously had a quit attempt using FDA-approved pharmacotherapy.
* Interest in reducing harms from tobacco use or quitting smoking

Exclusion Criteria

* Pregnant, breastfeeding, or trying to become pregnant.
* Household member currently enrolled in the study
* Planning to move out of the area within the next 7 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Biochemically-confirmed 7-day point prevalence abstinence from cigarettes on timeline followback | 11 Weeks
  Self-reported zero cigarettes in the past 7 days on timeline followback at Week 11 + expired carbon monoxide < 6 ppm

SECONDARY OUTCOMES:
Greater than 50% reduction in cigarette smoking | 11 Weeks
  Average reduction in the number of cigarettes smoked per day on 7-day timeline followback at Week 11 of at least 50% or greater compared to average baseline number of cigarettes smoked per day on 7 day timeline followback

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Smith, Principal Investigator — smithtra@musc.edu
Locations (1):
- Medical Univeristy of South Carolina, Charleston, South Carolina, United States